CLINICAL TRIAL: NCT02855970
Title: Development and Validation of a French Quality Of Life Scale Specific to Patients Who Have Suffered a Stroke
Brief Title: Validation of a French Quality of Life Questionnaire Adapted to Persons Who Have Suffered a Stroke
Acronym: QUALI STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Béjot 2014
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

ARMS (1):
- patient (Experimental)
  Interventions: Other: completion of a quality of life questionnaire

INTERVENTIONS:
Other: completion of a quality of life questionnaire

SUMMARY:
The aim of this work is to develop and validate a scale adapted to French cultural characteristics. It will be based on the SS-QoL scale and be simple and quick to use in everyday practice. It is not simply a translation. This transcultural adaptation requires linguistic and psychometric validation, by studying its validity, its reliability and its sensitivity to change, as though it were a new instrument. The investigators will then develop a short version by reducing the items and conduct a psychometric validation.

The translation and validation of a short French version of the SS-QoL scale will generate a reliable and sensitive, easy-to-use tool suitable for use in everyday practice.

The final objective is to use this tool as a principal judgement criterion in future therapeutic trials and in patients of the Dijon Stroke Registry to bring to light prognostic factors that affect quality of life so as to provide better management of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Patients following a first stroke (ischemic or non-traumatic cerebral parenchyma haemorrhage) followed at a consultation at Dijon CHU and included in the Dijon Stroke Registry cohort.
* Patients who have provided oral informed consent.
* Patients with national health insurance cover

Exclusion Criteria:

* History of symptomatic stroke.
* Meningeal haemorrhage.
* Severe visual or hearing handicap making it difficult to complete the questionnaire.
* Global severe aphasia and mutism making communication with the patient impossible-.
* Unable to read or speak French.
* Dementia prior to the stroke.
* Psychiatric disorders and dependence on alcohol/drugs.
* Bedridden before the stroke.
* Other comorbidities considered severe by the clinician and not related to the stroke that could have significantly impaired quality of life before the stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
responses to a quality of life questionnaire | Change compared with baseline score at Day 15, Day 60

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France